CLINICAL TRIAL: NCT02988947
Title: Effectiveness of a Psychological Intervention for the Control and Prevention of Pain and for Surgical Recovery in Patients Undergoing Total Knee Arthroplasty: a Prospective Randomized Controlled Trial
Brief Title: Effectiveness of a Psychological Intervention in Patients Undergoing Total Knee Arthroplasty
Acronym: PsInTKA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unavailability of the clinical team
Sponsor: University of Minho (Other)
Collaborators: Hospital de Braga (Other)
Responsible Party: Principal Investigator, Patrícia Ribeiro Pinto, Post-doctoral fellow, University of Minho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SFRH/BPD/103529/2014
Record Dates: First submitted 2016-08-09; First posted 2016-12-12 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Knee Arthroplasty, Total
Keywords: Knee Arthroplasty; Hypnosis; Pain Neuroscience Education; Pain; Catastrophizing; Optimism; Distress; Hope; Self-Efficacy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (PNE+HyP) (Experimental): Patients in this group will have 3 pre-surgical + 1 (or 2) reinforcement sessions in adition to standard TKA care. These interventions are based on Pain Neuroscience Education and Hypnosis and delivered according to standardized scripts.
  Interventions: Other: PNE+HyP
- Control Group (No Intervention): No intervention / Standard care

INTERVENTIONS:
Other: PNE+HyP — This is a combined PNE and Hypnosis psychological intervention. PNE is a cognitive based approach that highlights the biopsychosocial model of pain and focuses on neurophysiological and neurobiological processes and pain representation. Hypnosis aims at promoting pain control, increasing positive coping strategies, and targeting positive psychological variables.
  Arms: Intervention Group (PNE+HyP)

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a combined Pain Neuroscience Education (PNE) and Hypnosis (HyP) psychological intervention aiming at the control and prevention of pain and promotion of post-surgical recovery in patients undergoing Total Knee Arthroplasty

DETAILED DESCRIPTION:
This is a prospective Randomized Controlled Trial (RCT), comparing an experimental group (EG), submitted to a PNE/HyP based psychological intervention, and a control group (CG), submitted to usual treatment and care.

After recruitment and evaluation of inclusion/exclusion criteria, patients entering the study will sign the Informed Consent. Baseline evaluation is performed at 1 month pre-surgery and, afterwards, patients are randomly assigned to EG (PNE+Hyp plus usual care) or CG (usual care only). The EG will be submitted to 3 pre-surgical and 1 (or 2) post-surgical reinforcement sessions. At 1 month post-surgery, the intervention group will be subdivided and participants will be randomly assigned to receive a reinforcement session or no intervention at this point. The psychological intervention sessions are based on the educative principles of Pain Neuroscience Education and on Hypnosis strategies for the promotion of pain control, positive coping strategies and psychological variables.

Patients will be evaluated on 6 moments: T0 - baseline, 1 month pre surgery; T1 - post intervention/24h before surgery; T2 - 72h post-surgery; T3 - 1 month post surgery; T4 - 6 months post surgery; T5 - 12 months post intervention. Patients will fill in self report measures and perform physiological evaluation to analyse relevant bio-markers (salivary cortisol and α-amylase) that are related to stress levels and SNS functioning and translate the impact of psychological interventions on physiological parameters.

ELIGIBILITY:
Inclusion Criteria:

* Planned unilateral total knee arthroplasty due to gonarthrosis
* Giving consent to participate

Exclusion Criteria:

* Inability to write and read
* Cognitive deficit (assessed by MMSE)
* Revision TKA
* Bilateral TKA
* TKA for reasons other than gonarthrosis (fracture, malignancy or infection)
* Psychiatric or neurological deficit (e.g. Schizophrenia or Alzheimers')
* Diagnosis of rheumatoid arthritis, Psoriatic arthritis, Systemic lupus erythematosus, Anquilosant spondylitis or other severe disease
* Contralateral hip or knee arthroplasty in the previous 6 months
* Planned contralateral hip or knee arthroplasty in the next 6 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Pain intensity post-intervention as assessed by Numerical Rating Scale (NRS) and WOMAC | 24h before surgery
Pain intensity 72h post-surgery as assessed by NRS | 72h post-surgery
Pain intensity 1 month post-surgery as assessed by NRS and WOMAC | 1 month post-surgery
Pain intensity 6 months post-surgery as assessed by NRS and WOMAC | 6 months post-surgery
Pain intensity 12 months post-surgery as assessed by NRS and WOMAC | 12 months post-surgery

SECONDARY OUTCOMES:
Physical functioning post-intervention as assessed by WOMAC | 24h before surgery
Physical functioning 1 month post-surgery as assessed by WOMAC | 1 month post-surgery
Physical functioning 6 months post-surgery as assessed by WOMAC | 6 months post-surgery
Physical functioning 12 months post-surgery as assessed by WOMAC | 12 months post-surgery
Pain knowledge post-intervention as assessed by the Neurophisiology of Pain Questionnaire (NPQ) | 24h before surgery
Pain knowledge 1 month post-surgery as assessed by the NPQ | 1 month post-surgery
Pain knowledge 6 months post-surgery as assessed by NPQ | 6 months post-surgery
Pain knowledge 12 months post-surgery as assessed by NPQ | 12 months post-surgery
Emotional distress post-intervention as assessed by the Hospital Anxiety and Depression Scale (HADS) | 24h before surgery
Emotional distress 1 month post-surgery as assessed by HADS | 1 month post-surgery
Emotional distress 6 months post-surgery as assessed by HADS | 6 months post-surgery
Emotional distress 12 months post-surgery as assessed by HADS | 12 months post-surgery
Optimism post-intervention as assessed by the Life Orientation Test (LOT-R) | 24h before surgery
Optimism 1 month post-surgery as assessed by LOT | 1 month post-surgery
Optimism 6 months post-surgery as assessed by LOT-R | 6 months post-surgery
Optimism 12 months post-surgery as assessed LOT-R | 12 months post-surgery
Pain coping strategies post-intervention as assessed by the Coping Strategies Questionnaire (CSQ) | 24h before surgery
Pain coping strategies 1 month post-surgery as assessed by CSQ | 1 month post-surgery
Pain coping strategies at 6 months post-surgery as assessed by CSQ | 6 months post-surgery
Pain coping strategies at 12 months post-surgery as assessed by CSQ | 12 months post-surgery
Hope post-intervention as assessed by the Portuguese Hope Scale (Escala Sobre a Esperança - ESE) | 24h before surgery
Hope at 1 month post-surgery as assessed by ESE | 1 month post-surgery
Hope at 6 months post-surgery as assessed by ESE | 6 months post-surgery
Hope at 12 months post-surgery as assessed by ESE | 12 months post-surgery
Self-Efficacy post-intervention as assessed by the Self-Efficacy Scale developed for this study (KSESS) | 24h before surgery
Self-Efficacy at 1 month post-surgery as assessed by KSESS | 1 month post-surgery
Self-Efficacy at 6 months post-surgery as assessed by KSESS | 6 months post-surgery
Self-Efficacy at 12 months post-surgery as assessed by KSESS | 12 months post-surgery
Salivary cortisol levels post-intervention | 24h before surgery
Salivary cortisol levels 72h post-surgery | 72h post-surgery
Salivary cortisol levels at 1 month post-surgery | 1 month post-surgery
Salivary cortisol levels at 6 months post-surgery | 6 months post-surgery
Salivary cortisol levels at 12 months post-surgery | 12 months post-surgery
Salivary α-amylase levels post-intervention | 24h before surgery
Salivary α-amylase levels 72h post-surgery | 72h post-surgery
Salivary α-amylase levels at 1 month post-surgery | 1 month post- surgery
Salivary α-amylase at 6 months post-surgery | 6 months post-surgery
Salivary α-amylase at 12 months post-surgery | 12 months post-surgery
Inflammatory biomarkers | 24h before surgery
  IL-1β, IL-6, IL-10, TNFα, MCP-1, hs-CRP

CONTACTS AND LOCATIONS:
Locations (1):
- Life and Health Sciences Research Institute, Braga, Portugal

IPD SHARING:
Plan to Share IPD: No